CLINICAL TRIAL: NCT03732703
Title: Myeloma-Developing Regimens Using Genomics (MyDRUG) (Genomics Guided Multi-arm Trial of Targeted Agents Alone or in Combination With a Backbone Regimen)
Brief Title: Myeloma-Developing Regimens Using Genomics (MyDRUG)
Acronym: MyDRUG
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Multiple Myeloma Research Consortium (Network)
Collaborators: AbbVie (Industry); Celgene Corporation (Industry); Eli Lilly and Company (Industry); Genentech, Inc. (Industry); Janssen, LP (Industry); Takeda (Industry); GlaxoSmithKline (Industry); Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MyDRUG (MMRC-085)
Record Dates: First submitted 2018-10-29; First posted 2018-11-07 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Relapsed Refractory Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed Refractory; Multiple Myeloma Research Consortium (MMRC); Genomic Profile; My Drug; Multiple Myeloma Research Foundation
MeSH Terms: conditions — Multiple Myeloma | interventions — abemaciclib; Dexamethasone; ixazomib; pomalidomide; MLN2238; enasidenib; cobimetinib; erdafitinib; venetoclax; daratumumab; belantamab mafodotin; selinexor

STUDY DESIGN:
Intervention Model Description: Eight Arms with 38 patients per arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Sub-Protocol A1 (Experimental): Patients with CDK activating alteration receive Abemaciclib in combination with ixazomib, pomalidomide and dexamethasone (IPd)
  Interventions: Drug: Abemaciclib, dexamethasone, ixazomib, pomalidomide
- Sub-Protocol B1 (Experimental): Patients with IDH2 activating mutation receive Enasidenib in combination with ixazomib, pomalidomide and dexamethasone (IPd)
  Interventions: Drug: Enasidenib, dexamethasone, ixazomib, pomalidomide
- Sub-Protocol C1 (Experimental): Patients with the presence of RAF/RAS mutation receive Cobimetinib in combination with ixazomib, pomalidomide and dexamethasone (IPd)
  Interventions: Drug: Cobimetinib, dexamethasone, ixazomib, pomalidomide
- Sub-Protocol D1 (Experimental): Patients with presence of FGFR3 activating mutations receive Erdafitinib in combination with ixazomib, pomalidomide and dexamethasone (IPd)
  Interventions: Drug: Erdafitinib, dexamethasone, ixazomib, pomalidomide
- Sub-Protocol E1 (Experimental): Patients with t(11;14) translocation will be enrolled in arm E1 and randomized to the venetoclax or the IPd control arm. Patients with relapsed Multiple Myeloma will receive Venetoclax, Ixazomib, Pomalidomide and Dexamethasone every cycle. Each cycle is 28 days long.
  Interventions: Drug: Venetoclax, dexamethasone, ixazomib, pomalidomide
- Sub-Protocol Y1 (Experimental): Patients with Non-Actionable Genetic Abnormality receive Daratumumab in combination with ixazomib, pomalidomide and dexamethasone (IPd)
  Interventions: Drug: Daratumumab, dexamethasone, ixazomib, pomalidomide
- Sub-Protocol Y2 (Experimental): Patients with Non-Actionable Genetic Abnormality receive Belantamab mafodotin in combination with ixazomib, pomalidomide and dexamethasone (IPd)
  Interventions: Drug: Belantamab mafodotin, dexamethasone, ixazomib, pomalidomide
- Sub-Protocol Y3 (Experimental): Patients with Non-Actionable Genetic Abnormality receive Selinexor in combination with ixazomib, pomalidomide and dexamethasone (IPd)
  Interventions: Drug: Selinexor, dexamethasone, ixazomib, pomalidomide

INTERVENTIONS:
Drug: Abemaciclib, dexamethasone, ixazomib, pomalidomide — Patients with relapsed Multiple Myeloma will receive Abemaciclib and Dexamethasone for the first 2 cycles. Abemaciclib, Dexamethasone, Ixazomib and Pomalidomide from cycle 3 forward. Each cycle is 28 days long.
  Other Names: abemaciclib: Verzenio, LY2835219; ixazomib: Ninlaro, MLN2238; pomalidomide: Pomalyst
  Arms: Sub-Protocol A1
Drug: Enasidenib, dexamethasone, ixazomib, pomalidomide — Patients with relapsed Multiple Myeloma will receive Enasidenib and Dexamethasone for the first 2 cycles. Enasidenib, Dexamethasone, Ixazomib and Pomalidomide from cycle 3 forward. Each cycle is 28 days long.
  Other Names: enasidenib: AG221, IDHIFA; ixazomib: Ninlaro, MLN2238; pomalidomide: Pomalyst
  Arms: Sub-Protocol B1
Drug: Cobimetinib, dexamethasone, ixazomib, pomalidomide — Patients with relapsed Multiple Myeloma will receive Cobimetinib and Dexamethasone for the first 2 cycles. Cobimetinib, Dexamethasone, Ixazomib and Pomalidomide from cycle 3 forward. Each cycle is 28 days long.
  Other Names: cobimetinib: Cotellic, GDC-0973, RG7420; ixazomib: Ninlaro, MLN2238; pomalidomide: Pomalyst
  Arms: Sub-Protocol C1
Drug: Erdafitinib, dexamethasone, ixazomib, pomalidomide — Patients with relapsed Multiple Myeloma will receive Erdafitinib and Dexamethasone for the first 2 cycles. Erdafitinib, Dexamethasone, Ixazomib and Pomalidomide from cycle 3 forward. Each cycle is 28 days long.
  Other Names: erdafitinib: G-024, JNJ-42756493, JNJ-493; ixazomib: Ninlaro, MLN2238; pomalidomide: Pomalyst
  Arms: Sub-Protocol D1
Drug: Venetoclax, dexamethasone, ixazomib, pomalidomide — Patients with t(11;14) translocation will be enrolled in arm E1 and randomized to the venetoclax or the IPd control arm. Patients with relapsed Multiple Myeloma will receive Venetoclax, Ixazomib, Pomalidomide and Dexamethasone every cycle. Each cycle is 28 days long.
  Other Names: venetoclax: Venclexta: ABT-199; ixazomib: Ninlaro, MLN2238; pomalidomide: Pomalyst
  Arms: Sub-Protocol E1
Drug: Daratumumab, dexamethasone, ixazomib, pomalidomide — Patients with relapsed Multiple Myeloma will receive Daratumumab, Ixazomib, Pomalidomide and Dexamethasone every cycle. Each cycle is 28 days long.
  Other Names: daratumumab: Darzalex; ixazomib: Ninlaro, MLN2238; pomalidomide: Pomalyst
  Arms: Sub-Protocol Y1
Drug: Belantamab mafodotin, dexamethasone, ixazomib, pomalidomide — Patients with relapsed Multiple Myeloma will receive Belantamab mafodotin, Ixazomib, Pomalidomide and Dexamethasone every cycle. Each cycle is 28 days long.
  Other Names: Belantamab mafodotin: BLENREP, GSK2857916
  Arms: Sub-Protocol Y2
Drug: Selinexor, dexamethasone, ixazomib, pomalidomide — Patients with relapsed Multiple Myeloma will receive Selinexor, Ixazomib, Pomalidomide and Dexamethasone every cycle. Each cycle is 28 days long.
  Other Names: Selinexor: XPOVIO
  Arms: Sub-Protocol Y3

SUMMARY:
The MyDRUG study is a type of Precision Medicine trial to treat patients with drugs targeted to affect specific genes that are mutated as part of the disease. Mutations in genes can lead to uncontrolled cell growth and cancer. Patients with a greater than 25% mutation to any of the following genes; CDKN2C, FGFR3, KRAS, NRAS, BRAF V600E, IDH2 or T(11;14) can be enrolled to one of the treatment arms. These arms have treatments specifically directed to the mutated genes. Patients that do not have a greater than 25% mutation to the genes listed can be enrolled to a non-actionable treatment arm.

The genetic sequencing of the patient's tumor is required via enrollment to the MMRF002 study: Clinical-grade Molecular Profiling of Patients with Multiple Myeloma and Related Plasma Cell Malignancies. (NCT02884102).

DETAILED DESCRIPTION:
The study will enroll 228 patients enrolled to one of eight treatment arms. The study is open to patients relapsing with relapsed refractory multiple myeloma, who have

* received at least one prior but no more than 3 prior therapies
* exposed to both a PI and an IMiD
* had early relapse after initial treatment. Relapse is defined as the IMWG uniform response criteria (Kumar et al, 2016). Early relapse as defined by at least one of the following:

  1. Relapse within 3 years post autologous stem cell transplantation (ASCT) on maintenance, or 18 months if unmaintained
  2. Relapse within 18 months of initial non-ASCT based therapy

ELIGIBILITY:
Inclusion Criteria:

* Willing to be registered into the pomalidomide (POMALYST®) Risk Evaluation and Mitigation Strategy (REMS®) program
* Enrolled in the MMRF002 Molecular Profiling Protocol (NCT02884102) with report less than 120 days old
* Disease free of prior malignancies for ≥ 3 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, carcinoma "in situ" of the cervix or breast, or prostate cancer not requiring therapy
* High risk patients with relapsed refractory multiple myeloma (RRMM), who have:

  * received at least one prior but no more than 3 prior therapies
  * exposed to both a PI and an IMiD
  * had early relapse after initial treatment Early relapse as defined by at least one of the following: (Relapse is defined as the IMWG uniform response)

    1. Relapse within 3 years of initiation of induction chemo therapy for post autologous stem cell transplantation (ASCT) followed by maintenance, or 18 months if unmaintained after ASCT
    2. Within 18 months of initial non-ASCT based therapy
* Patients must have progressed after their most recent treatment and require therapy for myeloma
* Females of reproductive potential must have a negative pregnancy test at baseline, be non-lactating, and willing to adhere to scheduled pregnancy testing
* Females of reproductive potential and males must practice and acceptable method of birth control
* Laboratory values obtained ≤ 14 days prior to registration:

  * Absolute neutrophil count (ANC) ≥ 1000/ul
  * Hemoglobin (Hgb) ≥ 8 g/dl
  * Platelet (PLT) ≥ 75,000/ul
  * Total bilirubin <1.5 x upper limit of normal (ULN) or if total bilirubin is >1.5 x ULN, the direct bilirubin must be ≤ 2.0 mg/dL
  * Aspartate aminotransferase (AST) <3 x ULN
  * Creatinine Clearance ≥ 30 mL/min

Measurable disease of Multiple Myeloma (MM) as defined by at least one of the following:

* Serum monoclonal protein ≥ 0.5 g by protein electrophoresis
* ≥200 mg of monoclonal protein in the urine on 24-hour electrophoresis
* Serum immunoglobulin free light chain (FLC) ≥10 mg/dL AND abnormal serum immunoglobulin kappa to lambda FLC ratio
* Monoclonal bone marrow plasmacytosis ≥30% (evaluable disease)

  * Eastern Cooperative Oncology Group (ECOG) Performance Status 0, 1, or 2
  * Ability to take aspirin, warfarin, or low molecular weight heparin

Sub-Protocol Inclusion Criteria:

Refer to each respective Sub Protocol for additional inclusion criteria.

Exclusion Criteria:

Patients will be ineligible for this study if they meet any one of the following criteria:

* Aggressive multiple myeloma requiring immediate treatment as defined by:

  * Lactate dehydrogenase (LDH) > 2 times ULN
  * Presence of symptomatic extramedullary disease or central nervous system involvement
  * Hypercalcemia >11.5 mg/dl
  * Acute worsening of renal function (CrCl < 30 ml/min) directly related to myeloma relapse
  * Any neurological emergency related to myeloma
  * Clinical symptoms of hyperviscosity related to monoclonal protein
  * Involved serum free light chain > 100 mg/dL (1000 mg/L) in the setting of prior diagnosis of cast nephropathy
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days of enrolment
* Known hypersensitivity or development of erythema nodosum if characterized by a desquamating rash while taking thalidomide, lenalidomide, pomalidomide or similar drug. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of the agents
* Prior Ixazomib/Pomalidomide/Dexamethasone combination therapy
* Pregnant or breast-feeding females
* Serious medical or psychiatric illness, active alcoholism, or drug addiction that may hinder or confuse compliance, interfere in the completion of treatment per protocol, or follow-up evaluation
* Active hepatitis A, B or C viral infection or known human immunodeficiency virus (HIV) infection
* Concurrent symptomatic amyloidosis or plasma cell leukemia
* POEMS syndrome [plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes]
* Residual side effects to previous therapy > Grade 1 prior to initiation of therapy (Alopecia any grade and/or neuropathy Grade 2 without pain are permitted)
* Prior allogeneic or ASCT within 12 weeks of initiation of therapy. Prior allogeneic stem cell transplant with active graft-versus-host disease (GVHD)
* Prior experimental therapy within 14 days of protocol treatment or 5 half-lives of the investigational drug, whichever is longer
* Prior anticancer therapy within 14 days of initiation of protocol therapy (Dexamethasone/ 40mg/day) for a maximum of 4 days before screening is allowed
* Prior major surgical procedure or radiation therapy within 4 weeks of the initiation of therapy (this does not include limited course of radiation used for management of bone pain within 7 days of initiation of therapy).
* Known to have dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or Gastro Intestinal (GI) absorption of drugs administered orally
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months
* Other co-morbidity, which would interfere with patient's ability to participate in trial or that confounds the ability to interpret data from the study

Sub-Protocol Exclusion Criteria:

Refer to each respective Sub Protocol for additional exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate - Actionable Genetic Alteration | Patients will be evaluated monthly for response from the start of the study until the date of documented disease progression, assessed up to 2 years
  • To evaluate the overall response rate (ORR) with targeted agents used in combination with backbone regimen ixazomib, pomalidomide and dexamethasone (IPd) in patients with an actionable genetic alteration per the International Myeloma Working Group [IMWG] consensus criteria (Kumar et al, 2016)
Overall Response Rate - Non-Actionable Genetic Alteration | Patients will be evaluated monthly for response from the start of the study until the date of documented disease progression, assessed up to 2 years
  • To evaluate the ORR with agents used in combination with backbone (or IPd) regimen in patients with no actionable genetic alteration per IMWG consensus criteria (Kumar et al, 2016).

CONTACTS AND LOCATIONS:
Overall Officials: Hearn J Cho, M.D., Ph.D., Principal Investigator — Multiple Myeloma Research Consortium
Locations (16):
- United States (16):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - City of Hope, Duarte, California
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Karmanos Cancer Center, Detroit, Michigan
  - Mayo Clinic - Minnesota, Rochester, Minnesota
  - Washington University School of Medicine Division of Medical Oncology, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Ohio State University College of Medicine, Columbus, Ohio
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar S, Paiva B, Anderson KC, Durie B, Landgren O, Moreau P, Munshi N, Lonial S, Blade J, Mateos MV, Dimopoulos M, Kastritis E, Boccadoro M, Orlowski R, Goldschmidt H, Spencer A, Hou J, Chng WJ, Usmani SZ, Zamagni E, Shimizu K, Jagannath S, Johnsen HE, Terpos E, Reiman A, Kyle RA, Sonneveld P, Richardson PG, McCarthy P, Ludwig H, Chen W, Cavo M, Harousseau JL, Lentzsch S, Hillengass J, Palumbo A, Orfao A, Rajkumar SV, Miguel JS, Avet-Loiseau H. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. Lancet Oncol. 2016 Aug;17(8):e328-e346. doi: 10.1016/S1470-2045(16)30206-6. PMID 27511158